CLINICAL TRIAL: NCT02219958
Title: Evaluation of Quality of Care - Multi-disciplinary Risk Assessment and Management Programme for Patients With Hypertension, HA (QoC RAMP-HT)
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1685
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAMP-HT and Non-RAMP-HT

SUMMARY:
Hypertension (HT) is one of the major cause of morbidity and among the top 10 causes of deaths in Hong Kong in 2008 (Department of Health 2009). The Hospital Authority (HA) has initiated service improvement through introducing the risk assessment and management programme (RAMP) to improve the quality of care (QOC) for HT patients in general outpatient clinics (GOPC). The evaluation on the QOC is an essential part of the programme in order to inform future policy. The Department of Family Medicine and Primary Care (FMPC) of the University of Hong Kong (HKU) has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the RAMP programme is achieved. Each RAMP participating clinic and hospital will be invited to complete a structured evaluation questionnaire. The data of all patients who have enrolled into the RAMP for more than one year will be included in the evaluation on the process and outcomes of care.

One thousand two hundred and forty-eight age and disease matched control patients who have not been enrolled into the RAMP programme will be selected for the comparison in the outcomes of care. A hundred and thirty participants will be followed up by telephone to evaluate the effect of the programme in quality of life (QOL), patient enablement, and global rating of change in health condition at baseline and 6 months after enrolment. Data on the process of care will be retrieved from the HA medical records.

Main Outcome Measures: The primary outcomes are the proportion of participants who have received the criterion process of care, and achieved the target blood pressure levels.

Data Analysis: Descriptive statistics on proportions of centers or subjects meeting the QOC criteria will be calculated. The changes in the clinical and patient reported outcomes of RAMP subjects will be compared at 12, 24, 36 and 48 months will be compared by paired sample t-test. The clinical outcomes between RAMP subjects and control group will be compared by independent sample t-test or Chi-square test.

Results: The QOC of the RAMP programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified.

Conclusion: The results of this study will provide empirical evidence on whether the HA's RAMP programme can achieve improvement in QOC for HT patients. The information will be used to guide service planning and policy decision making.

ELIGIBILITY:
Inclusion Criteria:

* HT
* aged <80
* Suboptimal BP control (average systolic blood pressure (SBP) ≥ 140mmHg or average diastolic blood pressure (DBP) ≥ 90mmHg)

Exclusion Criteria:

* Patients will be excluded if they are unable to understand or communicate in Chinese language, or refuse to give consent.
* Patients will be excluded if they had prior history of diabetes and existing cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HT patients aged <80, without prior history of diabetes and existing cardiovascular diseases, with suboptimal BP control (average systolic blood pressure (SBP) ≥ 140mmHg or average diastolic blood pressure (DBP) ≥ 90mmHg) who were enrolled into RAMP-HT.
Sampling Method: Probability Sample
Enrollment: 2496 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clinics that have satisfied each of the structure criteria | Three years
  Final analysis will evaluate the period from August, 2012 to December, 2014.
The proportion of patients who have complied with the criterion process of care. | Three years
  Final analysis will evaluate the period from August, 2012 to December, 2014.
The proportion of patients who have achieved a BP level <140/90mmHg. | Three years
  Final analysis will evaluate the period from August, 2012 to December, 2014.

SECONDARY OUTCOMES:
LDL | Three years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 3 years.
BMI (Body Mass Index) | Three years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 3 years.
Occurrence of First Cardiovascular Complication | Three years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 3 years.
The change in SF-12v2 scores | Three years
  Baseline and 6-month/12-month/24-month/36-month after the first administration of questionnaire.
PEI (Patient Enablement Index) | Three years
  6-month/12-month/24-month/36-month after the first administration of questionnaire.
GRS (Global Rating of Change Scale) scores | Three years
  6-month/12-month/24-month/36-month after the first administration of questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong; Esther Y.T. Yu, MBBS, Principal Investigator — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong Island, Hong Kong

REFERENCES:
- [Result] Yu EY, Wan EY, Chan KH, Wong CK, Kwok RL, Fong DY, Lam CL. Evaluation of the quality of care of a multi-disciplinary Risk Factor Assessment and Management Programme for Hypertension (RAMP-HT). BMC Fam Pract. 2015 Jun 19;16:71. doi: 10.1186/s12875-015-0291-0. PMID 26088560
- [Derived] Yu EYT, Wan EYF, Mak IL, Chao DVK, Ko WWK, Leung M, Li YC, Liang J, Luk W, Wong MMY, Ha TKH, Chan AKC, Fong DYT, Lam CLK. Assessment of Hypertension Complications and Health Service Use 5 Years After Implementation of a Multicomponent Intervention. JAMA Netw Open. 2023 May 1;6(5):e2315064. doi: 10.1001/jamanetworkopen.2023.15064. PMID 37223900